CLINICAL TRIAL: NCT06521814
Title: Globus Reflect Tether - Humanitarian Use Device
Brief Title: Globus Reflect Tether - HUD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: This study was withdrawn prior to enrollment due to challenges in initiating the project. No participants were enrolled, and no data were collected. The study will not proceed further and is being formally closed.
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00132703
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Globus-tethering HUD patients (Experimental): The implantation of the REFLECT scoliosis tethering system in patients diagnosed with idiopathic scoliosis.
  Interventions: Procedure: REFLECT scoliosis correction system

INTERVENTIONS:
Procedure: REFLECT scoliosis correction system — (i.e. purpose of research) The Globus Reflect scoliosis correction system aims to provide curve correction for scoliosis patients who are still actively growing. Surgical correction is accomplished without spinal fusion, instead utilizing anterior vertebral body tethering. Reflect holds the convexity of the curve in place so that the concavity can grow, thereby harnessing the power of normal spine growth to correct the deformity.

SUMMARY:
The purpose of this device is to treat children and adolescents with scoliosis who have growth remaining. In patients with a curvature about the spine, Reflect holds the convexity of the curve in place so that the concavity can grow, thereby harnessing the power of normal spine growth to correct the deformity.

DETAILED DESCRIPTION:
The Globus Reflect scoliosis correction system aims to provide curve correction for scoliosis patients who are still actively growing. Surgical correction is accomplished without spinal fusion, instead utilizing anterior vertebral body tethering. This device received an HDE exemption from the FDA and requires MUSC IRB approval to be used.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally immature patients that require surgical treatment to obtain and maintain correction of progressive idiopathic scoliosis, with a major Cobb angle of 35 to 60 degrees whose osseous structure is dimensionally adequate to accommodate screw fixation, as determined by radiographic imaging.
* Patients should have failed bracing and/or be intolerant to brace wear.

Exclusion Criteria:

* Pregnancy (current)
* Prior spinal or chest surgery
* MRI abnormalities (including syrinx greater than 4mm, Chiari malformation, or tethered cord)
* Neuromuscular, thoracogenic, cardiogenic scoliosis, or any other non-idiopathic scoliosis
* Associated syndrome, including Marfan Disease or Neurofibromatosis
* Sanders stage greater than 4
* Thoracic curve less than 35 or greater than 60
* Lumbar curve greater than or equal to 35
* Unable or unwilling to firmly commit to returning for required follow-up visits
* Investigator judgement that the subject/family may not be a candidate for the intervention

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2025-11-01 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Cobb angles | Until patients reach the age of 18
  Decrease in cobb angles for patients who are actively still growing

CONTACTS AND LOCATIONS:
Overall Officials: Robert Murphy, Principal Investigator — Medical University of South Carolina